CLINICAL TRIAL: NCT00918606
Title: An Evaluation of the Pharmacokinetics and Safety of LIPO-102 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIPO-102-CL-01
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Subcutaneous Adipose Tissue Reduction

ARMS (1):
- LIPO-102 (Experimental)
  Interventions: Drug: LIPO-102

INTERVENTIONS:
Drug: LIPO-102 — LIPO-102

SUMMARY:
An Evaluation of the PK and Safety of LIPO-102 in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male and non pregnant female
* 18-55 years old
* Sufficient abdominal fat for injections
* Signed informed consent

Exclusion Criteria:

* Known hypersensitivity to study drugs
* Treatment with an investigational agent within 30 days before first dose

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety: Laboratory tests, medical exams | 4 weeks

SECONDARY OUTCOMES:
Pharmacokinetics | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore, Maryland, United States